CLINICAL TRIAL: NCT04112212
Title: Using Fluorescently Labeled Vedolizumab to Visualize Local Drug Distribution During Colonoscopy and Identify Mucosal Target Cells in Patients With Inflammatory Bowel Disease
Brief Title: Using Vedolizumab-800CW to Gain Insight Into Local Drug Distribution and Mucosal Target Cells in IBD Patients
Acronym: VISION
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: NL69572.042.19
Record Dates: First submitted 2019-09-25; First posted 2019-10-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Crohn Disease; Colitis, Ulcerative
Keywords: Fluorescence; Endoscopy; Vedolizumab-800CW
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 38 IBD patients were included in the study.
  1. Dose escalation, including 3 dose groups.
  2. Adding a blocking dose.
  3. Patients included after >14 weeks of therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No administration of vedolizumab-800CW (Other): Patients did not receive vedolizumab-800CW but underwent a Fluorescence molecular imaging procedure to serve as a control group and compare results with patients receiving the tracer
  Interventions: Other: Fluorescence molecular imaging procedure without prior administration of vedolizumab-800CW
- 4.5 mg vedolizumab-800CW group (Experimental): Patients received 4.5 mg vedolizumab-800CW and subsequently underwent a Fluorescence molecular imaging procedure
  Interventions: Drug: Fluorescence molecular imaging procedure using vedolizumab-800CW
- 15 mg vedolizumab-800CW group (Experimental): Patients received 15 mg vedolizumab-800CW and subsequently underwent a Fluorescence molecular imaging procedure
  Interventions: Drug: Fluorescence molecular imaging procedure using vedolizumab-800CW
- 75 mg vedolizumab + 15 mg vedolizumab-800CW group (Experimental): Patients received 75mg vedolizumab + 15 mg vedolizumab-800CW and subsequently underwent a Fluorescence molecular imaging procedure
  Interventions: Combination Product: Fluorescence molecular imaging procedure using vedolizumab-800CW with prior administration of unlabeled vedolizumab
- 300mg vedolizumab + 15mg vedolizumab-800CW group (Experimental): Patients received 300mg vedolizumab + 15 mg vedolizumab-800CW and subsequently underwent a Fluorescence molecular imaging procedure
  Interventions: Combination Product: Fluorescence molecular imaging procedure using vedolizumab-800CW with prior administration of unlabeled vedolizumab
- > 14 weeks of vedolizumab therapy + 15 mg vedolizumab-800CW group (Experimental): Patients received 300mg vedolizumab + 15 mg vedolizumab-800CW after >14 weeks vedolizumab therapy and subsequently underwent a Fluorescence molecular imaging procedure
  Interventions: Combination Product: Fluorescence molecular imaging procedure using vedolizumab-800CW with prior administration of unlabeled vedolizumab

INTERVENTIONS:
Drug: Fluorescence molecular imaging procedure using vedolizumab-800CW — First vedolizumab-800CW was administered intravenously. 2-4 days later a fluorescence molecular imaging procedure was performed to enable the visualization and detection of fluorescence signals.
  Arms: 15 mg vedolizumab-800CW group; 4.5 mg vedolizumab-800CW group
Other: Fluorescence molecular imaging procedure without prior administration of vedolizumab-800CW — Fluorescence molecular imaging was performed to enable the visualization and detection of fluorescence signals.
  Other Names: Control group
  Arms: No administration of vedolizumab-800CW
Combination Product: Fluorescence molecular imaging procedure using vedolizumab-800CW with prior administration of unlabeled vedolizumab — Patients on vedolizumab therapy received vedolizumab-800CW iv or patients first received an unlabeled dose of vedolizumab prior to the iv administration of vedolizumab-800CW. 2-4 days later a fluorescence molecular imaging procedure was performed to enable the visualization and detection of fluorescence signals.
  Arms: 300mg vedolizumab + 15mg vedolizumab-800CW group; 75 mg vedolizumab + 15 mg vedolizumab-800CW group; > 14 weeks of vedolizumab therapy + 15 mg vedolizumab-800CW group

SUMMARY:
Summary Vision Study

Crohn's Disease (CD) and Ulcerative Colitis (UC) are chronic idiopathic inflammatory bowel diseases (IBD). Vedolizumab is a humanized monoclonal antibody against α4β7 integrin, capable of blocking the migration of several immune cells across endothelium expressing MAdCAM-1. Vedolizumab is expensive and primary non-response is high in both CD and UC. Currently there are no predictors of response to vedolizumab and the actual mechanism of action has not yet been elucidated. To clarify the mechanism of action and gain better understanding of the high primary non-response rates, the University Medical Center Groningen (UMCG) developed a tracer fluorescently labeling vedolizumab. This study aims to gain insight into vedolizumab distribution and concentrations in the gut. The current study aims to identify the vedolizumab target cells in the inflamed gut mucosa using quantitative fluorescence molecular imaging (FMI). By gaining insight into local vedolizumab concentrations, drug distribution and by discovering target cells, we expect to gain insight into the mechanism of action of vedolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of IBD, or Ulcerative Colitis (UC) or Crohn's Disease (CD).
* Vedolizumab naïve and eligible for vedolizumab treatment.
* Age: 18 years or older.
* Written informed consent.

Exclusion Criteria:

* Prior vedolizumab treatment
* Vedolizumab contraindicated as therapy
* Pregnancy or breast feeding.
* Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Fluorescent signal in patients with IBD | After 18 months when study is completed.
  Quantification of fluorescent signal after a microdose of vedolizumab-800CW in inflamed and non-inflamed tissue in patients with IBD.

SECONDARY OUTCOMES:
Safety of Vedolizumab-800CW in patients with IBD | Interim analysis after 30 weeks (at least 5 patients included). Complete data of all patients when study is completed. Individual patients were followed up for 1 week after vedolizumab-800CW injection for AE's, SAE's and SUSAR's.
  Collect safety data of vedolizumab-800CW. Checking vital parameters and adverse events caused by the drug or intervention.
  Register and analyze all AE's, SAE's and SUSAR's caused by vedolizumab-800CW.
Semi-quantifying fluorescent signals in patients with IBD | Interim analysis after 30 weeks (at least 5 patients included). Complete data after 18 months when study is completed.
  Semi-quantification of the ex vivo mean fluorescent intensity signal of vedolizumab-800CW in biopsies by calculating the mean fluorescence intensity (FImean) of biopsy images generated with a fluorescence flatbed scanner
FMI ex vivo analysis to detect target cells | After 18 months when study is completed.
  To evaluate the degree of in vivo fluorescence intensity for differences in severity of inflammation and quantify the in vivo NIR fluorescent signal of vedolizumab-800CW using the spectroscopy probe and compare this to the ex vivo fluorescent signal levels in the biopsies taken (immunohistochemistry, RNA and DNA analysis).
Distribution of Vedolizumab in the inflamed gut | After 18 months when study is completed.
  To assess the (sub-)cellular location of vedolizumab-800CW microscopically.

CONTACTS AND LOCATIONS:
Overall Officials: W.B. Nagengast, MD, PhD, PharmD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tjalma JJJ, Koller M, Linssen MD, Hartmans E, de Jongh SJ, Jorritsma-Smit A, Karrenbeld A, de Vries EG, Kleibeuker JH, Pennings JP, Havenga K, Hemmer PH, Hospers GA, van Etten B, Ntziachristos V, van Dam GM, Robinson DJ, Nagengast WB. Quantitative fluorescence endoscopy: an innovative endoscopy approach to evaluate neoadjuvant treatment response in locally advanced rectal cancer. Gut. 2020 Mar;69(3):406-410. doi: 10.1136/gutjnl-2019-319755. Epub 2019 Sep 18. No abstract available. PMID 31533965
- [Background] Nagengast WB, Hartmans E, Garcia-Allende PB, Peters FTM, Linssen MD, Koch M, Koller M, Tjalma JJJ, Karrenbeld A, Jorritsma-Smit A, Kleibeuker JH, van Dam GM, Ntziachristos V. Near-infrared fluorescence molecular endoscopy detects dysplastic oesophageal lesions using topical and systemic tracer of vascular endothelial growth factor A. Gut. 2019 Jan;68(1):7-10. doi: 10.1136/gutjnl-2017-314953. Epub 2017 Dec 15. No abstract available. PMID 29247063
- [Derived] Gabriels RY, van der Waaij AM, Linssen MD, Dobosz M, Volkmer P, Jalal S, Robinson D, Hermoso MA, Lub-de Hooge MN, Festen EAM, Kats-Ugurlu G, Dijkstra G, Nagengast WB. Fluorescently labelled vedolizumab to visualise drug distribution and mucosal target cells in inflammatory bowel disease. Gut. 2024 Aug 8;73(9):1454-1463. doi: 10.1136/gutjnl-2023-331696. PMID 38580386